CLINICAL TRIAL: NCT03313817
Title: Pre and Post-arterial Recanalization Imaging of Central Retinal Artery Occlusions (CRAO)
Acronym: I-RECANAL
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2017_17
Record Dates: First submitted 2017-09-25; First posted 2017-10-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Retinal Artery Occlusion; Magnetic Resonance Imaging; Diagnosis; Etiology; Prognosis
MeSH Terms: conditions — Retinal Artery Occlusion; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Additional MRI sequences — Patients will be hospitalized for suspicion of CRAO. An "optimized" MRI will be performed with specific sequences: 3D T1 MSDE (Motion Sensitized Driven Equilibrium) "dark blood"; 3D Optimized diffusion centered on the optic nerves; 3D PD T1 after injection. A consultation of ophthalmology and a control MRI will be carried out one month after the CRAO. Again, specific sequences will be added: 3D T1 MSDE (Motion Sensitized Driven Equilibrium) "dark blood"; 3D Optimized diffusion centered on the optic nerves; DTI (Diffusion Tensor Imaging); 3D PD T1 after injection.

SUMMARY:
Central retinal artery occlusions (CRAO) are the equivalent of an ischemic stroke at the retinal level. They share the same risk factors and common pathology. The diagnosis of a CRAO is clinically based on the sudden occurrence of a decrease in deep visual acuity with fundamentally signs of reactive ischemia.

Small studies have highlighted the value of cerebral MRI (Magnetic Resonance Imaging) in CRAO with almost 25% of ischemic strokes found on diffusion sequences and the demonstration of a correlation between anomalies in diffusion sequence and the probability of a pathology with a high risk of recurrence (carotid stenosis or emboligenic cardiopathy). But there are usually few radiological signs that allow a direct positive diagnosis of CRAO, an etiologic diagnosis or a prognosis. This descriptive study will focus on CRAO at the diagnostic and post-treatment phases in the short and medium term, in order to (i) identify imaging etiologic signs of CRAO with specific sequences from a 3 Tesla MRI, (ii) identify positive diagnostic signs of CRAO with the same specific sequences, (iii) correlate these signs with the visual prognosis one month after the CRAO.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* CRAO (onset of symptoms ≤ 48 hours)
* Consent to participate in the study

Exclusion Criteria:

- Contraindications to 3 Tesla MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized for CRAO ≤ 48 hours.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement of the ophthalmic artery | Baseline
  Binary variable (yes/no)
Presence of a thrombus | Baseline
  Binary variable (yes/no)
Presence of an arterial stenosis of the supra aortic trunks | Baseline
  Binary variable (yes/no)
Hypersignal of the ophthalmic artery in diffusion | Baseline
  Binary variable (yes/no)
Restriction of the apparent diffusion coefficient (ADC) at the optic nerve level and at the papilla level | Baseline
  Binary variable (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No